CLINICAL TRIAL: NCT02897609
Title: Clinical Evaluation of Beta-Lacta ™ Test in Urinary Infections
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BETA-LACTA
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2016-09

CONDITIONS: Urinary Infection
Keywords: Beta-lactamine; β-lactamine
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A simple questionary filled

SUMMARY:
3rd generation cephalosporins (C3G) are the antibiotics recommended in probabilistic in most enteric infections in France including pyelonephritis and bacteraemia.

However, the prevalence of resistance of Enterobacteriaceae including E. coli to C3G is continuously increasing for several years. In 2012, in France, the proportion of E. resistant or intermediate coli categorized to C3G is 10 to 25% (EARSS data).

Antibiotics not adapted early in severe sepsis is responsible for worse prognosis for patients in terms of morbidity and mortality and unnecessary prolongation of the DMS.

At St. Joseph's Hospital on enterobacteria levels of resistance to C3G is 15.4%.

To avoid overuse of carbapenems for probabilistic antibiotic and to quickly prescribe antibiotics adapted to the resistance of the bacteria, it is interesting to use a rapid test for detection of resistance to C3G.

The Lacta ™ test could be used in this indication. This is a rapid test diagnostic orientation detecting hydrolysis of a substrate (chromogenic cephalosporin) by the enzymatic action of ESBL, cAMP-type cephalosporinases and carbapenemases. This test was initially marketed for rapid detection of resistance to C3G enterobacteria from isolated bacterial colonies in culture.

DETAILED DESCRIPTION:
Main objective / secondary:

The investigators propose to conduct a study with a double objective:

1. To assess the analytical performance and its positioning relative to all the tests available to us in urine samples,
2. To evaluate prospectively the clinical impact test in urinary infections

Expected results and prospects:

This study will define the performance and limitations of this test in the most difficult situations (low number of bacteria / ml, haematic urine, ...) and will specify its indications and its place among all other tests before implanting it in our routine, as appropriate.

The clinical impact study will provide medical and economic analysis data including shortening time to adapt antibiotic therapies and put in septic isolation to argue the implementation of this test routinely.

ELIGIBILITY:
Inclusion Criteria:

* Patients may have a urinary infection ESBLE
* Patients accepting the use of their result for analysis.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients may have a urinary infection ESBLE
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the relevance between antibiotic susceptibility and the antibiotic chosen,with phone questionary | Hour 48
  The biologist advise, as usual, the physician about the antibiotic to choose at H0 according to the result of Beta Lacta™Test. After the first result given, the biologist ask, at hour 48,the physician about the antibiotic chosen and determine the relevance according to the antibiotic susceptibility.
  The answer can be yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Alban LE MONNIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mizrahi A, Naouri D, Hobson C, Amzalag J, Pilmis B, Couzigou C, Ganansia O, Le Monnier A. Impact of the beta-lacta test on the management of urinary tract infections at the emergency department. Infect Dis (Lond). 2021 Jan;53(1):52-60. doi: 10.1080/23744235.2020.1822543. Epub 2020 Sep 22. PMID 32960659